CLINICAL TRIAL: NCT06295133
Title: Determining the Influence of a Stress Management Intervention on Medical Students Levels of Psychophysiological Stress and Satisfaction.
Brief Title: Preventive Remediation of Stress for Optimal MEdical StudentS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PROMESS - STRESS
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Health Behavior; Health-Related Behavior; Stress
Keywords: Health; Student; Curriculum; Behaviour; Medical; Stress
MeSH Terms: conditions — Health Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: All volunteers will receive a stress management intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress intervention (Experimental): One arm : all volunteers will receive a stress management intervention.
  Interventions: Behavioral: Stress

INTERVENTIONS:
Behavioral: Stress — The stress management intervention will consist of three individual sessions, each lasting one hour, with approximately 15 days between each session. The sessions will be scheduled as follow: week 5 and 6 (session 1), week 7 and 8 (session 2), week 9, 10, and 11 (session 3). During these sessions, subjective and objective indicators of stress will be recorded to assess the progress of each student.

SUMMARY:
Medical students are subjected to a high competitive pressure throughout their curriculum. High levels of stress are associated with a deterioration in quality of life and learning abilities.

Our field surveys conducted in 2022 and 2023 at the Lyon Est Medical School revealed that second-cycle students presented a high level of stress. It is expected that these feelings significantly degrade their quality of life as well as their health. Furthermore, a local survey reported that one in two medical students had experienced at least one depressive episode, and one in three had already had suicidal thoughts during their curriculum.

Thus, it would become crucial for medical students to manage stressful situations and reduce stress levels during their studies.

The PROMESS - STRESS project aims to offer solutions to students to reduce their stress levels during their medical studies. It responds to a demand expressed by students : our previous field study showed that 45% of fourth-year students declared being "very interested" and/or "interested" in following a intervention aimed at stress reduction. An early knowledge of stress remediation tools would allow students to quickly acquire the necessary tools to cope with stressful situations they will encounter during their training and their life as future physicians. The objective of this study is to determine the influence of a stress management intervention on medical students levels of psychophysiological stress and satisfaction.

DETAILED DESCRIPTION:
Our project aims to support future healthcare professionals to adopt health-promoting behaviors during their studies in a preventive approach. This support will be provided through an intervention of stress management during their curriculum. Specifically, 4th and 5th-year students of the Faculty of Medicine of Lyon Est will have the opportunity to participate in the PROMESS STRESS project. 45 voluntaries will follow a preventive program based on stress management. This intervention will span 11 weeks. At the end of this period, we expect improvements in both subjective and objective indicators of stress.

METHODS.

PRE-INTERVENTION. Week 1. Participants will undergo a two-hour session, during which, they will complete questionnaires on stress. We will also record Heart Rate Variability (HRV).

INTERVENTION. From week 5 to week 11. The stress management intervention will consist of three individual sessions, each lasting one hour, with approximately 15 days between each session. Each session includes individual interviews between a stress expert and the participant (i.e. student).

The sessions will be scheduled as follow: week 5 and 6 (session 1), week 7 and 8 (session 2), week 9, 10, and 11 (session 3). During the interview, the expert realizes an initial assessment of student stress levels and gives personalized goals to student. Subsequent sessions follow the same structure.

ELIGIBILITY:
Inclusion Criteria:

* Being a 4th-year or a 5th-year medical student at the Faculty of Medicine Lyon East during the academic year 2023-2024.
* Having read the information note.
* Having signed the written consent.

Exclusion Criteria:

* No exclusion criteria will be applied.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Perceived level of stress : Evolution of the score obtained at the Perceived Stress Scale (PSS). | From week 5 to week 11.
  The students level of stress will be assessed through the PSS questionnaire ranging from 0 (none) to 40 (extreme). One score is assessed and can be classified as low, moderate and elevated stress. The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).

SECONDARY OUTCOMES:
Scale of Holmes and Rahe : score obtained at the Holmes and Rahe Questionnaire Inventory. | Week 1 (Pre-intervention).
  Quantity of stressors met by the students during the last years. One score is assessed and can be classified as low, medium and high risk of health degradation. This measure will be done during the pre-interventional period at week 1.
Big-5 : scores obtained at the Big-5 questionnaire. | Week 1 (Pre-intervention).
  The students personality traits (i.e. agreeableness, openness, consciousness, extraversion, neuroticism) will be assessed through the questionnaire each score ranges from one to five. This measure will be done during the pre-interventional period at week 1.
Coping strategies : scores obtained at the Brief Cope Inventory (BCI). | Week 1 (Pre-intervention).
  The students coping strategies (social support, active resolution, positive thinking, and avoidance) will be assessed through the BCI questionnaire, each score ranging from 1 to 4; a high score indicating that the behaviour was highly engaged. This measure will be done during the pre-interventional period at week 1.
Perceived level of stress : score obtained at the Perceived Stress Scale | Week 1 (Pre-intervention).
  The students level of stress will be assessed through the PSS questionnaire ranging from 0 (none) to 40 (extreme). One score is assessed and can be classified as low, moderate and elevated stress.This measure will be done during the pre-interventional period at week 1.
Heart rate variability (HRV) marker: cardiac coherence score during the pre-intervention. | Week 1 (Pre-intervention).
  The students basal level of physiological stress will be assessed through the cardiac coherence score, an HRV marker. This measure will be done during the pre-interventional period at week 1.
Heart rate variability (HRV) marker: SDNN during the pre-intervention. | Week 1 (Pre-intervention).
  The students basal level of physiological stress will be assessed through the SDNN score, an HRV marker. SDNN is the standard deviation of the inter-beat-intervals (IBI) measured in ms, NN means "normal" beats, i.e, removing abnormal or false beats. This measure will be done during the pre-interventional period at week 1.
Heart rate variability (HRV) marker: RMSSD during the pre-intervention. | Week 1 (Pre-intervention).
  The students basal level of physiological stress will be assessed through the RMSSD, an HRV marker. RMSSD is the most commonly measured form of HRV, it calculates the difference between successive inter-beat-intervals (IBI) in ms, squares these values and takes the root of the mean.This measure will be done during the pre-interventional period at week 1.
Heart rate variability (HRV) marker: Low frequency / High frequency ratio (LF/HF) during the pre-intervention. | Week 1 (Pre-intervention).
  The students basal level of physiological stress will be assessed through the LF/HF ratio, an HRV marker. HF. The HF band is typically correlated with RMSSD and NN50, lower HF power is associated with stress and anxiety. It is primarily associated with activity in the parasympathetic nervous system.
  LF. The LF band is typically associated with the sympathetic nervous system and the HF/LF ratio is often used as a measure of sympathetic-parasympathetic balance in the nervous system.
  This measure will be done during the pre-interventional period at week 1.
Heart rate variability (HRV) marker: pnn50% during the pre-intervention. | Week 1 (Pre-intervention).
  The students basal level of physiological stress will be assessed through the pnn50%, an HRV marker. NN50 is the Number of pairs of successive intervals that differ by greater than 50ms. And pNN50 which is more typically used is the proportion of NN50 over all N-N intervals in a sample, expressed as a percentage.This measure will be done during the pre-interventional period at week 1.
Coping strategies : Evolution in scores obtained at the Brief Cope Inventory (BCI). | From week 5 to week 11.
  The students coping strategies (social support, active resolution, positive thinking, and avoidance) will be assessed through the BCI questionnaire each score will range from 1 to 4; a high score indicating that the behaviour was highly engaged. The measure will be done every session, session 1 (week 5-6) and session 2 (week 7-8), session 2 and session 3 (week 9,10,11).
Heart rate variability (HRV) marker: Evolution in cardiac coherence score during the intervention. | From week 5 to week 11.
  The students level of physiological stress will be assessed through the cardiac coherence, an HRV marker. The measure will be done every session, session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Heart rate variability (HRV) marker: Evolution in SDNN score during the intervention. | From week 5 to week 11.
  The students level of physiological stress will be assessed through the SDNN, an HRV marker.The measure will be done every session, session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Heart rate variability (HRV) marker: Evolution in RMSSD score during the intervention. | From week 5 to week 11.
  The students level of physiological stress will be assessed through the RMSSD, an HRV marker.
  The measure will be done every session, session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Heart rate variability (HRV) marker: Evolution in LF/HF ratio during the intervention. | From week 5 to week 25.
  The students level of physiological stress will be assessed through the LF/HF ratio, an HRV marker. The measure will be done every session, session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Heart rate variability (HRV) marker: Evolution in pnn50% score during the intervention. | From week 5 to week 11.
  The students level of physiological stress will be assessed through the pnn50%, an HRV marker. The measure will be done every session, session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - stressors quantity - Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived quantity of stressors | From week 5 to week 11.
  The students quantity of stressors will be assessed on a 100-mm Visual Analogue Scale (VAS: "In the past two weeks, how many stressful situations have you encountered?") ranging from 0 (maximum/extreme) to 100 (zero). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - stress quantity - Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of stress. | From week 5 to week 11.
  The students level of stress will be assessed on a 100-mm Visual Analogue Scale (VAS: "In the past two weeks, how would you characterize your stress level?") ranging from 0 (maximum stress) to 100 (no stress at all). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - stress quality: Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the emotional valence associated with the stress level. | From week 5 to week 11.
  The emotional valence associated of the students stress level will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your stress?") ranging from 0 (very negative feeling) to 100 (very positive feeling).The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - stress coping: Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the management of stressful situations. | From week 5 to week 11.
  The students management of stressful situations will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how did you manage your stressful situations?") ranging from 0 (very bad stress coping) to 100 (excellent stress coping). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Advices given by the expert. Score obtained on a Likert scale ranging from 1 to 5 characterizing the nature of the advices given by the expert. | From week 5 to week 11.
  Following each session, the expert reported if he/she has given during the interview a specific advice according to a pre-established list. For each pre-established advice, he/she has to report if :
  1. He/she didn't mention this
  2. He/she mentioned this but didn't directly advise it
  3. He/she mentioned this and recommended it
  4. He/she had set this in the goals
  5. The student was already doing it (positive reinforcement) The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert estimation of student's achievements. Score obtained on a Likert scale ranging from 1 to 3 accessing if the expert estimates that the student has achieve the goals previously set. | From week 5 to week 11.
  The expert evaluates, from 0 to 3 (i.e. 0 : not achieved at all, 1: slightly achieved, 2: fairly well achieved, 3: well achieved) if he/she estimates that the student has achieve the goals previously set.
  The measure will be done at session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert satisfaction. Scores obtained on a Likert scale ranging from 1 to 5 accessing the expert's satisfaction of his/her intervention. | From week 5 to week 11.
  The perceived level of the expert satisfaction ("Are you satisfied with the session you just realized?") will be accessed on a likert scale ranging from 1 (not at all satisfied) to 5 (very satisfied). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert level of comfort. Score assessing the expert comfort levels in participant relationships on a likert scale ranging from 1 to 5. | From week 5 to week 11.
  The perceived level of expert comfort of the relationship with the student ("How comfortable did you feel with the student?") will be accessed on a likert scale ranging from 1 (not at all comfortable) to 5 (very comfortable). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert estimation of the overall student's achievements. Score obtained on a Likert scale ranging from 1 to 5 accessing the expert's level of satisfaction on the student's progress. | Week 9-10-11
  The level of expert satisfaction of the student's progress ("Are you satisfied with the student's progress during the all intervention?") will be accessed on a likert scale ranging from 1 (not at all satisfied) to 5 (very satisfied). This measure will be done at the session 3, i.e. approximately at week 9,11,10.
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the all intervention. | Week 9-10-11
  The composite score will be the mean of two sub-scores :
  1. An intervention specific score : mean of the score obtained at the 100-mm Visual Analogue Scale (VAS: "Do you think the intervention has helped you to decrease your stress level?") ranging from 0 (absolutely not) to 100 (completely) and score obtained at the 100-mm Visual Analogue Scale (VAS :"Do you think the intervention allowed you to better manage the stressful events you encountered?") ranging from 0 (absolutely not) to 100 (completely).
  2. An intervention general score : mean of the score obtained at the 100-mm Visual Analogue Scale (VAS : "Do you think the proposed goals were suitable for your daily life?") ranging from 0 (absolutely not) to 100 (completely) and the score obtained at the 100-mm Visual Analogue Scale (VAS: "Do you think you can sustain the habit changes?") ranging from 0 (absolutely not) to 100 (completely).
  This measure will be done at the session 3, i.e. approximately at week 9,11,10.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Schlatter, Dr., Principal Investigator — RESHAPE U1290 INSERM UCBL-LYON 1 Rockfeller, Lyon France.
Locations (1):
- RESHAPE, Lyon, France

REFERENCES:
- [Derived] Metais A, Omarjee M, Valero B, Gleich A, Mekki A, Henry A, Duclos A, Lilot M, Rode G, Schlatter S. Determining the influence of an intervention of stress management on medical students' levels of psychophysiological stress: the protocol of the PROMESS-Stress clinical trial. BMC Med Educ. 2025 Feb 11;25(1):225. doi: 10.1186/s12909-024-06344-8. PMID 39934759